CLINICAL TRIAL: NCT02710500
Title: Phase I Intramuscular Gene Transfer Clinical Trial for Dysferlin Deficiency Delivering the Dysferlin Gene by AAVrh74
Brief Title: rAAVrh74.MHCK7.DYSF.DV for Treatment of Dysferlinopathies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB15-00669
Record Dates: First submitted 2016-02-11; First posted 2016-03-16 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Dysferlinopathy
Keywords: LGMD2B; Limb Girdle Muscular Dystrophy; Miyoshi; Gene Transfer; Dysferlin
MeSH Terms: conditions — Dysferlinopathy; Limb-girdle muscular dystrophy, type 2B; Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Low Dose) (Experimental): Three (n=3) dysferlin deficiency subjects will receive bilateral injections with one extensor digitorum brevis muscle (EDB) receiving the rAAVrh74.MHCK7.DYSF.DV and the other side receiving saline alone.Subjects will receive a total dose of 2 x 10^12 in one muscle.
  Intervention Drug: rAAVrh.MHCK7.DYSF.DV
  Interventions: Drug: rAAVrh74.MHCK7.DYSF.DV
- Cohort 2 (High Dose) (Experimental): Three (n=3) dysferlin deficiency subjects will receive bilateral injections with one extensor digitorum brevis muscle (EDB) receiving the rAAVrh74.MHCK7.DYSF.DV and the other side receiving saline alone.Subjects will receive a total dose of 6 x 10^12 vg in one muscle.
  Intervention Drug: rAAVrh74.MHCK7.DYSF.DV
  Interventions: Drug: rAAVrh74.MHCK7.DYSF.DV

INTERVENTIONS:
Drug: rAAVrh74.MHCK7.DYSF.DV — Biological/Vaccine: rAAVrh74.MHCK7.DYSF.DV Recombinant adeno-associated virus carrying a dysferlin transgene under control of a muscle specific MHCK7 promoter.

SUMMARY:
The proposed clinical trial is a double-blind, randomized controlled study with direct intramuscular injection of rAAVrh.74.MHCK7.DYSF.DV gene vector to the extensor digitorum brevis muscle (EDB). Two cohorts of subjects with dysferlin deficiency, each with proven mutations will undergo gene transfer. A minimum of three subjects will be enrolled into each cohort.

DETAILED DESCRIPTION:
This is a phase I safety and tolerability study with a direct intramuscular injection of rAAVrh.74.MHCK7.DYSF.DV transferred to the extensor digitorum brevis muscle (EDB). The study is designed as a randomized, controlled, dose escalation trial with one EDB receiving the rAAVrh.74.MHCK7.DYSF.DV and the other side receiving saline alone. It will follow the previously safe and effective IM gene transfer to EDB for LGMD2D.2, 3 The first cohort, inclusive of three Dysferlinopathy subjects, will receive a gene transfer total dose of 2 x 10^12 vector genomes. Muscle biopsies will be performed at Day 45 (two subjects) and Day 90 (one subject). If there are no safety concerns, three additional subjects will be enrolled and receive an escalated dose at 6 X 10^12 vg (total dose). Muscle biopsies in the second cohort will be performed at Day 90 (one subject) and Day 180 (two subjects). This protocol design gives us a maximum period of observation ranging from 6 weeks to 6 months to capture both transient and delayed gene expression, and to recognize sustained expression.

ELIGIBILITY:
Inclusion Criteria:

* Must be Non-ambulant (cannot walk 10 meters in ≤ 30 sec) and age 18 years or older
* Established mutations of the dysferlin gene on both alleles
* Impaired muscle function but with sufficient muscle preservation to ensure muscle transfection based on magnetic resonance image of the EDB showing sufficient muscle preservation to permit transfection
* Willingness of sexually active subjects with reproductive capacity to practice reliable method of contraception (If appropriate), during the first six months after gene transfer (females) or until two negative sperm samples are obtained post gene transfer (males).

Exclusion Criteria:

* Active viral infection based on clinical observations or serological evidence of HIV, or Hepatitis A, B or C infection
* The presence of a Dysferlin mutations without weakness or loss of function
* Symptoms or signs of cardiomyopathy, including:
* Dyspnea on exertion, pedal edema, shortness of breath upon lying flat, or rales at the base of the lungs
* Echocardiogram with ejection fraction below 40%
* Diagnosis of (or ongoing treatment for) an autoimmune disease
* Persistent leukopenia or leukocytosis (WBC ≤ 3.5 K/µL or ≥ 20.0 K/µL) or an absolute neutrophil count < 1.5K/µL
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer
* Pregnancy
* AAVrh74 or AAV8 binding antibody titers > 1:50 as determined by ELISA immunoassay
* Abnormal laboratory values in the clinically significant range in the table below, based upon normal values in the Nationwide Children's Hospital Laboratory: GGT, Total Bilirubin, Cystatine, Hemoglobin, White Blood Cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Determination of safety based on the development of unacceptable toxicity | 2 Years
  Defined as the occurrence of any one Grade III or higher, unanticipated, treatment-related toxicity

SECONDARY OUTCOMES:
Number of participants showing dysferlin protein expression in muscle tissue | 2 Years
  More than 3 fold increase in dysferlin protein expression in muscle compared to control side by western blot or more than 30% increase in dysferlin-expressing fibers
  Dysferlin protein expression as demonstrated with N -terminal anti-dysferlin antibodies will be quantified using BioQuant
Leukocyte marker counts including CD45, CD3, CD4, CD8, and MAC 387. | 2 Years
  Number of CD4+ cells/ mm2 area; Number of CD8+ cells/ mm2 area; Number of muscle fibers expressing MHCI staining / mm2 area; Number of muscle fibers expressing MHCII staining / mm2 area
Binding antibodies counts and ELISpot counts to both rAAVrh74 capsid and dysferlin protein. | 2 Years
  AAVrh74 or AAV8 binding antibody titers > 1:50 as determined by ELISA immunoassay
Number of inflammatory cells in muscle | 2 Years
  Number of inflammatory cells per mm2 area

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Mendell, MD, Principal Investigator — Director, Center for Gene Therapy
Locations (1):
- Nationwide Children's Hosptial, Columbus, Ohio, United States

REFERENCES:
- [Background] Sondergaard PC, Griffin DA, Pozsgai ER, Johnson RW, Grose WE, Heller KN, Shontz KM, Montgomery CL, Liu J, Clark KR, Sahenk Z, Mendell JR, Rodino-Klapac LR. AAV.Dysferlin Overlap Vectors Restore Function in Dysferlinopathy Animal Models. Ann Clin Transl Neurol. 2015 Mar;2(3):256-70. doi: 10.1002/acn3.172. Epub 2015 Jan 20. PMID 25815352
- [Background] Grose WE, Clark KR, Griffin D, Malik V, Shontz KM, Montgomery CL, Lewis S, Brown RH Jr, Janssen PM, Mendell JR, Rodino-Klapac LR. Homologous recombination mediates functional recovery of dysferlin deficiency following AAV5 gene transfer. PLoS One. 2012;7(6):e39233. doi: 10.1371/journal.pone.0039233. Epub 2012 Jun 15. PMID 22720081
- See also: Center for Gene Therapy, The Research Institute at Nationwide Children's Hospital — http://www.nationwidechildrens.org/center-for-gene-therapy